CLINICAL TRIAL: NCT02799212
Title: Evaluation of Postoperative Ascites After Somatostatin Infusion Following Hepatectomy for Hepatocellular Carcinoma: Multicenter Randomized Double-blind Placebo Controlled Trial (SOMAPROTECT01)
Brief Title: Evaluation of Postoperative Ascites After Somatostatin Infusion Following Hepatectomy for Hepatocellular Carcinoma
Acronym: SOMAPROTECT01
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 69HCL16_0129; 2016-004230-20 (EudraCT Number)
Record Dates: First submitted 2016-06-09; First posted 2016-06-14 (Estimated); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; Hepatectomy; Ascites; Somatostatin
MeSH Terms: conditions — Carcinoma, Hepatocellular; Ascites

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): postoperative somatostatin infusion during 5 days at 6mg/day, followed by one day at 3mg/day
  Interventions: Drug: somatostatin infusion
- Control group (Placebo Comparator): Placebo infusion (50ml of 0.9% NaCl/day) during 6 days
  Interventions: Drug: placebo infusion

INTERVENTIONS:
Drug: somatostatin infusion — postoperative somatostatin infusion during 5 days at 6mg/day, followed by one day at 3mg/day.
  Arms: Experimental group
Drug: placebo infusion — Placebo infusion (50ml of 0.9% NaCl/day) during 6 days.
  Arms: Control group

SUMMARY:
Most patients undergoing hepatectomy for hepatocellular carcinoma (HCC) suffer from underlying liver disease and are exposed to the risk of postoperative ascites, with subsequent morbidity, liver and renal failure, the need for specific treatments and prolonged hospital stay. Postoperative ascites is favored by an imbalance between portal venous inflow and the diminished hepatic venous outflow. Finding a reversible, non-invasive method for modulating the portal inflow would be of interest: it could be used temporarily during the early postoperative course to prevent acute portal hypertension. Somatostatin, a well-known drug already used in several indications, may limit the risk of postoperative ascites and liver failure by decreasing portal pressure after hepatectomy for HCC in patients with underlying liver disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with HCC diagnosed by histology or by imaging findings according to the Barcelona Clinic Liver Cancer Group
* Patients with a single or multiple HCCs deemed to be resectable with a curative intent at the preoperative evaluation
* Patients for whom an indication for hepatectomy has been decided and approved by multidisciplinary board:
* by laparotomy
* by coelioscopy with resection of at least 2 liver segments
* Patients with any underlying liver disease with or without proven cirrhosis, regarding histological features (including F2-F3-F4 fibrosis with or without cirrhosis) or with other evidence of a diseased liver if no biopsy has been performed preoperatively (dysmorphic liver or evidence of portal hypertension at imaging findings, oesophageal varices at endoscopy)
* Age ≥ 18 years
* Patients with ability to understand and sign a written inform consent form
* Patients who will be available for follow-up

Exclusion Criteria:

* Patients participating in another interventional research in progress or including an exclusion period still in progress at pre-inclusion (except interventional research with minimal risks and constraints that do not interfere with the judgement criteria of the study according to the judgement of the coordinating investigator).
* Patients with evidence of a healthy liver at biopsy

Disease-associated non-inclusion criteria include:

* Another histologic type of hepatic tumor besides HCC
* Distant extra-hepatic metastases, including peritoneal carcinomatosis
* The existence of complete portal thrombosis of the main portal trunk

Operative technique-associated non-inclusion criteria include:

- Indication of coelioscopy with resection of less than 2 liver segments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
presence of postoperative ascites during the postoperative course | Day 90
  The presence of postoperative ascites during the postoperative course defined by:
  * ≥500 ml / 24h of fluid in the drains during at least 3 days. Or
  * ascites requiring puncture or drainage

SECONDARY OUTCOMES:
Duration of ascites | Day 90
  Number of days with ≥ 500ml / 24h of ascites
Volume of ascites | Day 90
  Total ascites volume
postoperative morbidity | Day 90
  Postoperative morbidity according to Dindo-Clavien
Postoperative morbidity on Liver failure | Day 90
  Presence and severity of hepatic failure according to International Study Group of Liver Surgery (ISGLS)
Postoperative morbidity on Renal failure | Day 90
  Presence and severity of renal failure according to RIFLE scale (RIFLE: Risk, Injury, Failure, Loss of kidney function, and End-stage kidney disease)

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - APHP - Hôpital Beaujon, Clichy
  - CHRU Lille - Hopital Huriez, Lille
  - Hospices Civils de Lyon - Hôpital de la Croix Rousse, Lyon
  - APHM - Hôpital de la Timone, Marseille
  - CHU de Bordeaux - Hôpital Haut Lévèque, Pessac
  - CHU Rennes - Hôpital Pontchaillou, Rennes
  - CHU de Toulouse - Hopital Rangueil, Toulouse

REFERENCES:
- [Background] Mohkam K, Rayar M, Adam JP, Muscari F, Rode A, Merle P, Pradat P, Bauler S, Delfour I, Chiche L, Ducerf C, Boudjema K, Lesurtel M, Laurent C, Mabrut JY. Evaluation of postoperative ascites after somatostatin infusion following hepatectomy for hepatocellular carcinoma by laparotomy: a multicenter randomized double-blind controlled trial (SOMAPROTECT). BMC Cancer. 2018 Aug 23;18(1):844. doi: 10.1186/s12885-018-4667-0. PMID 30139340